CLINICAL TRIAL: NCT04634981
Title: Does the Mode of Anesthesia Affect the Feto-maternal Outcome in Category-1 Caesarean Section: A Prospective Non-randomized Study Comparing Spinal Versus General Anesthesia
Brief Title: Does the Mode of Anesthesia Affect the Feto-maternal Outcome in Category-1 Caesarean Section
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Samar Rafik Mohamed Amin, lecturer of anesthesia and surgical ICU, Benha University
Other Study IDs: REC-FOMBU 000048
Record Dates: First submitted 2020-10-23; First posted 2020-11-18 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2020-11

CONDITIONS: Anesthesia; Adverse Effect; Newborn Morbidity
Keywords: emergency cesarean section; general anesthesia; spinal; feto-maternal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group general anesthesia (G): patients will positioned with pelvic wedge on operating table and preoxygenated. Then rapid sequence induction with precalculated doses of propofol (2 mg/kg) and rocuronium (0.9 mg/kg) will followed by endotracheal intubation. After delivery of the baby, fentanyl will be administered. Later, anesthesia will be maintained with isoflurane (1%).
  Interventions: Procedure: anesthesia of emergency cesarean section
- Group Spinal anesthesia (S): all parturients will co-loaded with 500 ml of colloid solution. In the left lateral position, the patients' back will be cleaned with povidone iodine. In the meantime, the spinal anesthetic drug and local anesthetic drug will be prepared. After wiping povidone iodine with alcohol, a rapid single shot of 2.5 ml of 0.5% hyperbaric bupivacaine will be administered intrathecally using 22 G spinal needle. Oxygen will be administered using simple face mask till the delivery of the baby.
  Interventions: Procedure: anesthesia of emergency cesarean section

INTERVENTIONS:
Procedure: anesthesia of emergency cesarean section — compare General versus spinal anesthesia

SUMMARY:
Spinal anesthesia (SA) has become the standard technique in elective cesarean section (CS) as it results in less maternal and neonatal morbidity than general anesthesia (GA) (Grade-A recommendation, NICE). For women requiring emergency CS, rapid sequence general anesthesia (RSGA) is commonly used because this technique is faster to perform than SA. Though several randomized trials have compared the maternal and fetal outcome between these two anesthetic techniques, the studies with respect to category 1 CS (emergent conditions that hold immediate threat to life of the woman or fetus) are limited.

DETAILED DESCRIPTION:
Full term pregnant females will be included in this study. They will be allocated into two groups:

(Group G): will receive rapid sequence general anesthesia, and (Group S): will receive spinal anesthesia. After preoperative assessment and investigations by the attending anesthesiologist, the decision of the anesthetic approach will be decided by the attending anesthesiologist according to indications for CS.

Before induction of anesthesia intravenous (IV) ranitidine 50 mg will be administered after establishing an IV access. On the operating table, vital signs will be monitored for all parturients throughout the surgery according to the standard departmental protocol.

fetal well being will be assessed after delivery by using 1 minute and 5 min APGAR score and umbilical cord PH . in addition to maternal vital signs intra-operative then follow up any complications that may occur to the mother post-operative.

ELIGIBILITY:
following inclusion criteria:

* American Society of Anesthesiologists physical status (ASA) < III
* Age 18-40 year
* Gestational age>37 weeks
* Emergency cesarean delivery
* Singleton pregnancy

The exclusion criteria are:

* Twin pregnancy
* Disagreement of the patient
* Neurological impairment
* Congenital fetal abnormality
* body mass index > 40 kg/m2; and
* Sensitivity to any of the drugs used during the emergency CS.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — full term pregnant females
Study Population: full term pregnant women from 18-40 years old
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
APGAR score | 5 minutes after delivery
  Apgar score is a method for assessment of neonatal well-being after birth (0-3: severely depressed, 4-6: moderately depressed, 7-10: excellent condition)

SECONDARY OUTCOMES:
decision-to-delivery interval (DDI) | from decision to operate till delivery of the baby
  the interval in minutes from the time of the decision by obstetrician to the time of delivery of the baby
Umbilical cord PH | immediately after delivery
  Arterial blood gases from umbilical cord artery were used to assess newborn's acid-base status
Occurrence of maternal complications postoperative | from recovery from anesthesia up to 24 hours postoperative
  all mother were followed for any postoperative complications related to the anesthesia.
Neonatal ICU admission | from delivery of the baby up to 24 hour postoperative
  Admission to the NICU in percentage of the total participants.
Length of hospital stay | up to 1 month
  Length of stay (LOS) is the duration of a single episode of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Samar Rafik Mohamed Amin, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided